CLINICAL TRIAL: NCT03814005
Title: A Phase 1/1b Study of Pevonedistat in Combination With Select Standard of Care Agents in Patients With Higher-Risk Myelodysplastic Syndromes, Chronic Myelomonocytic Leukemia, Acute Myelogenous Leukemia, or Advanced Solid Tumors With Severe Renal Impairment or Mild or Moderate Hepatic Impairment
Brief Title: A Study of Pevonedistat in People With Blood Cancers or Solid Tumors With Kidney or Liver Problems
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: Pevonedistat-1016; U1111-1220-1396 (Other: WHO); 2018-004049-17 (EudraCT Number)
Record Dates: First submitted 2019-01-21; First posted 2019-01-23 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Acute; Renal Insufficiency; Liver Disease; Neoplasms
Keywords: Drug therapy
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Acute; Renal Insufficiency; Liver Diseases; Neoplasms | interventions — Azacitidine; pevonedistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Control Arm (Experimental): Pevonedistat 20 milligram per square meter (mg/m^2), infusion, intravenously, once, on Day 1 of Part A in participants with hematologic malignancies, followed by a washout period of approximately 4 to 7 days, further followed by azacitidine 75 mg/m^2, injection, subcutaneously in Cycle 1 or subcutaneously or intravenously in Cycle 2 and subsequent cycles, once on Day 1 through Day 7 or Day 1 through Day 5, and on Days 8 and 9 in combination with pevonedistat 20 mg/m^2, infusion, intravenously, once, on Days 1, 3, and 5 in each 28-day treatment cycle in participants with hematologic malignancies until symptomatic deterioration or PD, discontinuation for any reason, study stopped by the sponsor, or up to 12 cycles.
  Interventions: Drug: Azacitidine; Drug: Pevonedistat
- Renal Arm (Experimental): Pevonedistat 20 mg/m^2, infusion, intravenously, once, on Day 1 of Part A in participants with hematologic malignancies, followed by a washout period of approximately 4 to 7 days, further followed by azacitidine 75 mg/m^2, injection, subcutaneously in Cycle 1 or subcutaneously or intravenously in Cycle 2 and subsequent cycles, once on Day 1 through Day 7 or Day 1 through Day 5, and on Days 8-9 in combination with a starting dose of pevonedistat 10 mg/m^2 to a maximum dose of pevonedistat 15 mg/m^2, infusion, intravenously, once, on Days 1, 3, and 5 in each 28-day treatment cycle in participants with hematologic malignancies until symptomatic deterioration or PD, discontinuation for any reason, study stopped by the sponsor, or up to 12 cycles.
  Interventions: Drug: Azacitidine; Drug: Pevonedistat
- Mild Hepatic Arm (Experimental): Pevonedistat 20 mg/m^2, infusion, intravenously, once, on Day 1 of Part A in participants with hematologic malignancies, followed by a washout period of approximately 4 to 7 days, further followed by azacitidine 75 mg/m^2, injection, subcutaneously in Cycle 1 or subcutaneously or intravenously in Cycle 2 and subsequent cycles, once on Day 1 through Day 7 or Day 1 through Day 5, and on Days 8 and 9 in combination with a starting dose of pevonedistat 10 mg/m^2 to a maximum dose of pevonedistat 20 mg/m^2, infusion, intravenously, once, on Days 1, 3, and 5 in each 28-day treatment cycle in participants with hematologic malignancies until symptomatic deterioration or PD, discontinuation for any reason, study stopped by the sponsor, or up to 12 cycles.
  Interventions: Drug: Azacitidine; Drug: Pevonedistat

INTERVENTIONS:
Drug: Azacitidine — Azacitidine subcutaneous or intravenous injection.
Drug: Pevonedistat — Pevonedistat intravenous infusion.
  Other Names: TAK-924 and MLN4924

SUMMARY:
Pevonedistat is a medicine to treat people with blood cancers or solid tumors.

The main aim of the study is to learn about the levels of pevonedistat in the blood of participants with blood cancers or solid tumors, who also have severe kidney problems or mild to moderate liver problems. The information from this study will be used to work out the best dose of pevonedistat to give people with these conditions in future studies. At the first visit, the study doctor will check who can take part in the study.

This study is in 2 parts: A and B.

Part A Participants will be placed into 1 of 4 treatment groups depending on how severe their kidney and liver problems are. All participants will receive 1 dose of pevonedistat as a slow injection in their vein (infusion). Then, the study doctors will check the levels of pevonedistat in the blood of the participants for 3 days after the infusion. They will also check if the participants have any side effects from pevonedistat.

Participants will be asked to continue to Part B. Those who don't want to continue will visit the clinic 30 days later for a final check-up.

Part B Participants who agree to participate into Part B will receive an infusion of pevonedistat on specific days during a 21-day or 28-day cycle. The cycle time will depend on what type of cancer the participants have. Participants will also be treated with standard of care medicines for their kidney and liver problems during this time. In the first cycle, the study doctors will also check the levels of pevonedistat in the blood and urine of participants for 3 days after the infusion. Participants will continue with cycles of treatment together with standard of care medicines until their condition gets worse or they have too many side effects from the treatment.

When treatment has finished, participants will visit the clinic 10 days later for a final check-up.

DETAILED DESCRIPTION:
The drug being tested in this study is called pevonedistat. The study will characterize the PK of pevonedistat, assess the safety, and determine the dose of pevonedistat, in combination with azacitidine, docetaxel OR paclitaxel plus carboplatin in participants with higher-risk myelodysplastic syndromes (HRMDS), myelodysplastic syndromes (MDS), chronic myelomonocytic leukemia (CMML), acute myelogenous leukemia (AML), or advanced solid tumors who also have severe renal impairment or mild or moderate hepatic impairment.

The study will enroll approximately 42 participants. Participants with solid tumors or hematologic malignancies will be assigned to one of the four treatment groups on the basis of their renal and hepatic function:

* Control Arm (Normal Renal and Hepatic Function)
* Renal Arm (Severe Renal Impairment)
* Mild Hepatic Arm (Mild Hepatic Impairment)
* Moderate Hepatic Arm (Moderate Hepatic Impairment)

The study will be conducted in 2 parts: Part A and Part B. Part A will include single dose administration of pevonedistat. Eligible participants from Part A who will opt to continue treatment in Part B will be treated with pevonedistat in combination with standard of care (SOC) agents (azacitidine, docetaxel OR paclitaxel plus carboplatin) in Part B.

Intrapatient dose escalation of pevonedistat and SOC agents will be based on the safety data from Cycle 1 of Part B as mentioned below:

* In renal arm (severe renal impairment ) based on the safety data from Cycle 1 of Part B, pevonedistat may be increased to 15 mg/m^2 on Days 1, 3, and 5 of Cycle 2 Part B and in subsequent Cycles, to a maximum dose of 25 mg/m^2. Participants may be eligible for intrapatient dose escalation to paclitaxel 175 mg/m^2 in Cycle 2 or beyond if the lower dose is well tolerated. Intrapatient dose escalation of carboplatin to AUC5 will be allowed if treatment with AUC4 in Cycle 1 of Part B is safe and tolerable.
* In mild hepatic arm (mild hepatic impairment), the starting dose for pevonedistat and azacitidine in combination are not escalated in the cohort. Intrapatient dose escalation of carboplatin to AUC5 will be allowed if treatment with AUC4 in Cycle 1 of Part B is safe and tolerable.
* In moderate hepatic arm (moderate hepatic impairment) based on the safety data from Cycle 1 of Part B, pevonedistat may be increased to 15 mg/m^2 on Days 1, 3, and 5 of Cycle 2 Part B and in subsequent Cycles, to a maximum dose of 20 mg/m^2. Intrapatient dose escalation of carboplatin to AUC5 will be allowed if treatment with AUC4 in Cycle 1 of Part B is safe and tolerable.

This multi-center trial will be conducted in the United States and Spain. The overall time to participate in this study is approximately 3.5 years. Participants will attend end of the study visit 30 days after the last dose of study drug or before the start of subsequent therapy, if that occurs sooner for safety follow up.

ELIGIBILITY:
Inclusion Criteria:

All participants:

1. Has expected survival of at least 3 months from the date of enrollment in the study.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
3. Has recovered (that is, Grade <=1 toxicity) from the reversible effects of prior anticancer therapy.
4. Prothrombin time (PT) and activated partial thromboplastin time (aPTT) <=1.5 * upper limit of the normal range (ULN) at screening or within 7 days before the first dose of study drug.
5. Suitable venous access for the study-required blood sampling (that is, PK sampling).

   For hematologic malignancies:
6. Previously untreated hematologic malignancies not suitable for induction therapy.
7. Morphologically confirmed diagnosis of MDS or nonproliferative CMML (that is, with white blood cell [WBC] <13,000 /mcL) at the study entry, based on one of the following:

   French-American-British (FAB) Classifications:
   * Refractory anemia with excess blasts (RAEB), defined as having 5% to 20% myeloblasts in the bone marrow.
   * CMML with 10% to 19% myeloblasts in the bone marrow and/or 5% to 19% blasts in the blood.

   OR

   World Health Organization (WHO) Classifications:
   * RAEB-1, defined as having 5% to 9% myeloblasts in the bone marrow.
   * RAEB-2, defined as having 10% to 19% myeloblasts in the bone marrow and/or 5% to 19% blasts in the blood.
   * CMML-2, defined as having 10% to 19% myeloblasts in the bone marrow and/or 5% to 19% blasts in the blood.
   * CMML-1 (although CMML-1 is defined as having <10% myeloblasts in the bone marrow and/or <5% blasts in the blood, these participants may enroll only if bone marrow blasts >=5%).
8. With MDS or CMML and must also have one of the following Prognostic Risk Categories, based on the Revised International Prognostic Scoring System (IPSS-R):

   * Very high (>6 points).
   * High (>4.5-6 points).
   * Intermediate (>3-4.5 points): a participant determined to be in the Intermediate Prognostic Risk Category is only allowable in the setting of >=5% bone marrow myeloblasts.
9. With WHO-defined AML at study entry, including leukemia secondary to prior chemotherapy or resulting from an antecedent hematologic disorder, have failed to achieve CR or have relapsed after prior therapy and are not candidates for potentially curative treatment.
10. With relapsed or refractory MDS, have previously been treated with an hypomethylating agent.
11. Laboratory value requirements per study arms are:

    * Estimated glomerular filtration rate (eGFR) (milliliter per minute per 1.73 square meter [mL/min/1.73^m]) >=90 (Control arm), <30 (Renal arm) , >=60 (Mild and Moderate hepatic arm).
    * Total Bilirubin <= ULN (Control arm), <= ULN (Renal arm), ULN <Bilirubin <=1.5 * ULN (not secondary to transfusions) (Mild hepatic arm) and 1.5 * ULN <bilirubin <=3.0 * ULN (not secondary to transfusions) (Moderate hepatic arm).
    * Alanine aminotransferase (ALT) <= ULN (Control arm), <=2.5 * ULN (Renal arm) and any value (for mild and moderate hepatic arm).

    For advanced solid tumors:
12. Have a histologically or cytologically confirmed metastatic or locally advanced solid tumor that is appropriate for treatment with pevonedistat in combination with either docetaxel or carboplatin plus paclitaxel in Part B of this study, or have progressed despite standard therapy, or whom conventional therapy is not considered effective.
13. Computerized tomography (CT) scan or magnetic resonance imaging (MRI) of the chest, abdomen, and pelvis within 28 days of the first dose of the study drug.
14. Laboratory value requirements per study arms are:

    * eGFR (mL/min/1.73m^2) <30 (Renal arm) and >=60 (mild and moderate hepatic arm).
    * Total bilirubin <=ULN (Renal arm), ULN <bilirubin <=1.5 * ULN (Mild hepatic arm) and 1.5 * ULN <bilirubin <=3.0 * ULN (Moderate hepatic arm).
    * ALT <=1.5 * ULN (for participants who receive pevonedistat plus docetaxel only) or <=2.5 * ULN (for participants who receive pevonedistat plus carboplatin plus paclitaxel only) (Renal arm) and any value (Mild and Moderate hepatic arm).

Exclusion Criteria:

All participants:-

1. With end-stage renal disease requiring hemodialysis.
2. Has Gilbert syndrome.
3. Has active uncontrolled infection or severe infectious disease, such as severe pneumonia, meningitis, or septicemia. Prophylactic treatment with antibiotics is allowed.
4. Has life-threatening illness unrelated to cancer.
5. Known human immunodeficiency virus (HIV) seropositive.
6. Treatment with strong cytochrome P450 (CYP)3A inducers within 14 days before the first dose of pevonedistat.
7. Has left ventricular ejection fraction (LVEF) <50% within 6 months prior to study enrollment. If a result within this time frame is unavailable, LVEF must be determined by echocardiography or multigated acquisition scan at screening.
8. Has severe uncontrolled ventricular arrhythmias or torsade de pointes; electrocardiographic evidence of acute ischemia or active conduction system abnormalities; or clinically significant arrhythmia (as an example, well-controlled atrial fibrillation would not be an exclusion whereas uncontrolled atrial fibrillation would be an exclusion).
9. Has severe symptomatic pulmonary hypertension requiring pharmacologic therapy or participants with chronic respiratory disease that requires continuous oxygen.

   For hematologic malignancies:
10. Has acute promyelocytic leukemia as diagnosed by morphologic examination of bone marrow, by fluorescent in situ hybridization or cytogenetics of peripheral blood or bone marrow, or by other accepted analysis.
11. With AML with a WBC count >=50,000/mcL. Participants who are cytoreduced with leukapheresis or with hydroxyurea may be enrolled if they otherwise meet the eligibility criteria.
12. With either clinical evidence of or history of central nervous system (CNS) involvement by AML.
13. With hematologic malignancies, PT or aPTT >1.5 * ULN or active uncontrolled coagulopathy or bleeding disorder. Participants therapeutically anticoagulated with warfarin, direct thrombin inhibitors, direct factor Xa inhibitors, or heparin are excluded from enrollment.

    For advanced solid tumors:
14. Has prior treatment with radiation therapy involving >=25% of the hematopoietically active bone marrow.
15. Has CNS metastasis, except for participants who have received prior treatment (radiation or resection) and have stable CNS disease (example: stable MRI, no steroid requirement).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2022-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (8):
- United States (2):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
- Spain (6):
  - ICO lHospitalet Hospital Duran i Reynals, LHospitalet de Llobregat, Barcelona
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital de San Pedro de Alcantara, Cáceres
  - C.H. Regional Reina Sofia, Córdoba
  - Complejo Asistencial Universitario de Salamanca H. Clinico, Salamanca
  - Hospital Universitario Virgen del Rocio - PPDS, Seville

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b603a4db2bf003ab4a2d1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 5 investigative sites in United States and Spain from 10 July 2019 to 19 April 2022.
Pre-assignment Details: Participants with myelodysplastic syndromes (MDS), and acute myelogenous leukemia (AML) who also had severe renal impairment or mild hepatic impairment were enrolled in this study to receive single dose of pevonedistat in Part A followed by a wash out period and pevonedistat in combination with standard of care agent in Part B. No participants with chronic myelomonocytic leukemia (CMML) and solid tumors were enrolled in this study.
Groups:
- Control Arm: Pevonedistat 20 mg/m^2, infusion, intravenously (IV), once, on Day 1 of Part A in participants with hematologic malignancies, followed by a washout period of approximately 4 to 7 days. Following Part A participants received azacitidine 75 mg/m^2, injection, subcutaneously (SC) in Cycle 1 or SC or IV in Cycle 2 and subsequent cycles, once on Day 1 through Day 7 or Day 1 through Day 5, and on Days 8 and 9 in combination with pevonedistat 20 mg/m^2, infusion, IV, once, on Days 1, 3, and 5 in each 28-day treatment cycle in participants with hematologic malignancies in Part B until symptomatic deterioration or PD, discontinuation for any reason, study stopped by the sponsor, or up to 12 cycles.
- Renal Arm: Pevonedistat 20 mg/m^2, infusion, intravenously, once, on Day 1 of Part A in participants with hematologic malignancies, followed by a washout period of approximately 4 to 7 days. Following Part A participants received azacitidine 75 mg/m^2, injection, subcutaneously in Cycle 1 or subcutaneously or intravenously in Cycle 2 and subsequent cycles, once on Day 1 through Day 7 or Day 1 through Day 5, and on Days 8-9 in combination with a starting dose of pevonedistat 10 mg/m^2 to a maximum dose of pevonedistat 15 mg/m^2, infusion, intravenously, once, on Days 1, 3, and 5 in each 28-day treatment cycle in participants with hematologic malignancies in Part B until symptomatic deterioration or PD, discontinuation for any reason, study stopped by the sponsor, or up to 12 cycles.
- Mild Hepatic Arm: Pevonedistat 20 mg/m^2, infusion, intravenously, once, on Day 1 of Part A in participants with hematologic malignancies, followed by a washout period of approximately 4 to 7 days. Following Part A participants received azacitidine 75 mg/m^2, injection, subcutaneously in Cycle 1 or subcutaneously or intravenously in Cycle 2 and subsequent cycles, once on Day 1 through Day 7 or Day 1 through Day 5, and on Days 8 and 9 in combination with a starting dose of pevonedistat 10 mg/m^2 to a maximum dose of pevonedistat 20 mg/m^2, infusion, intravenously, once, on Days 1, 3, and 5 in each 28-day treatment cycle in participants with hematologic malignancies until symptomatic deterioration or PD, discontinuation for any reason, study stopped by the sponsor, or up to 12 cycles.
Period: Part A: Day 1 to Day 4
Arm/Group | Control Arm | Renal Arm | Mild Hepatic Arm
Started | 10 | 4 | 3
Response-evaluable Population (Response-evaluable population included participants who received at least 1 dose of study drug, had a baseline disease assessment, and had at least 1 postbaseline disease assessment to analyze response.) | 8 | 1 | 2
Completed | 10 | 4 | 3
Not Completed | 0 | 0 | 0
Period: Washout Period : Day 4 to Day 7
Arm/Group | Control Arm | Renal Arm | Mild Hepatic Arm
Started | 10 | 4 | 3
Completed | 10 | 4 | 3
Not Completed | 0 | 0 | 0
Period: Part B: Day 8 to Day 343
Arm/Group | Control Arm | Renal Arm | Mild Hepatic Arm
Started | 10 | 4 | 3
Completed | 0 | 0 | 0
Not Completed | 10 | 4 | 3
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 3
Not completed — Progressive Disease | 4 | 2 | 0
Not completed — Unsatisfactory Therapeutic Response | 2 | 0 | 0
Not completed — Symptomatic Deterioration | 1 | 2 | 0
Not completed — Reason not Specified | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of study drug.
Groups:
- Control Arm: Pevonedistat 20 milligram per square meter (mg/m^2), infusion, intravenously (IV), once, on Day 1 of Part A in participants with hematologic malignancies, followed by a washout period of approximately 4 to 7 days. Following Part A participants received azacitidine 75 mg/m^2, injection, subcutaneously (SC) in Cycle 1 or SC or IV in Cycle 2 and subsequent cycles, once on Day 1 through Day 7 or Day 1 through Day 5, and on Days 8 and 9 in combination with pevonedistat 20 mg/m^2, infusion, IV, once, on Days 1, 3, and 5 in each 28-day treatment cycle in participants with hematologic malignancies in Part B until symptomatic deterioration or PD, discontinuation for any reason, study stopped by the sponsor, or up to 12 cycles.
- Total: Total of all reporting groups
Arm/Group | Control Arm | Renal Arm | Mild Hepatic Arm | Total
Number analyzed (Participants) | 10 | 4 | 3 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.1 (11.75) | 71.5 (6.86) | 79.7 (3.06) | 72.1 (10.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 2
  Male | 10 | 3 | 2 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 4 | 3 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 8 | 4 | 2 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 3 | 2 | 11
  Spain | 4 | 1 | 1 | 6
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 170.3 (5.99) | 175.0 (11.13) | 170.2 (22.00) | 171.4 (10.40)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 75.0 (7.77) | 74.5 (14.21) | 71.7 (19.43) | 74.3 (10.98)

OUTCOME MEASURES:

1. Primary Outcome: Part A, AUC∞: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity for Pevonedistat Following a Single Dose
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: Pharmacokinetic (PK) population included all participants who had sufficient dosing in Part A and Part B Cycle 1, had sufficient concentration-time data to permit reliable estimation of PK parameters, and who had not received any excluded concomitant medications through the completion of Part A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter(h*ng/mL)
Groups:
- Part A: Control Arm: Pevonedistat 20 mg/m^2: Pevonedistat 20 mg/m^2, infusion, IV, once, on Day 1 of Part A in participants with normal renal and hepatic function with hematologic malignancies (MDS and AML).
- Part A: Renal Arm: Pevonedistat 20 mg/m^2: Pevonedistat 20 mg/m^2, infusion, IV, once, on Day 1 of Part A in participants with severe renal impairment with hematologic malignancies (MDS and AML).
- Part A: Mild Hepatic Arm: Pevonedistat 20 mg/m^2: Pevonedistat 20 mg/m^2, infusion, IV, once, on Day 1 of Part A in participants with mild hepatic impairment with and hematologic malignancies (MDS and AML).
Arm/Group | Part A: Control Arm: Pevonedistat 20 mg/m^2 | Part A: Renal Arm: Pevonedistat 20 mg/m^2 | Part A: Mild Hepatic Arm: Pevonedistat 20 mg/m^2
Number analyzed (Participants) | 10 | 4 | 3
hour*nanogram per milliliter(h*ng/mL) | 1168.616 (69.4811) | 1293.467 (22.0685) | 1050.553 (69.4854)

2. Primary Outcome: Part A, AUClast: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration for Pevonedistat Following a Single Dose
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: PK population included all participants who had sufficient dosing in Part A and Part B Cycle 1, had sufficient concentration-time data to permit reliable estimation of PK parameters, and who had not received any excluded concomitant medications through the completion of Part A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Part A: Mild Hepatic Arm: Pevonedistat 20 mg/m^2: Pevonedistat 20 mg/m^2, infusion, IV, once, on Day 1 of Part A in participants with mild hepatic impairment with hematologic malignancies (MDS and AML).
Arm/Group | Part A: Control Arm: Pevonedistat 20 mg/m^2 | Part A: Renal Arm: Pevonedistat 20 mg/m^2 | Part A: Mild Hepatic Arm: Pevonedistat 20 mg/m^2
Number analyzed (Participants) | 10 | 4 | 3
h*ng/mL | 1120.759 (73.3956) | 1267.523 (22.1528) | 1020.344 (71.9314)

3. Primary Outcome: Part A, Cmax: Maximum Observed Plasma Concentration for Pevonedistat Following a Single Dose
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter(ng/mL)
Arm/Group | Part A: Control Arm: Pevonedistat 20 mg/m^2 | Part A: Renal Arm: Pevonedistat 20 mg/m^2 | Part A: Mild Hepatic Arm: Pevonedistat 20 mg/m^2
Number analyzed (Participants) | 10 | 4 | 3
nanograms per milliliter(ng/mL) | 262.9 (188.54) | 180.2 (37.66) | 148.9 (30.09)

4. Secondary Outcome: Parts A and B, t1/2z: Terminal Disposition Phase Half-life for Pevonedistat Following Single and Multiple Dose
Time Frame: Part A: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose; Part B: Cycle 1 Day 3 pre-dose and at multiple time points (up to 48 hours) post-dose (Cycle length= 28 days)
Population: PK population included all participants who had sufficient dosing in Part A and Part B Cycle 1, had sufficient concentration-time data to permit reliable estimation of PK parameters, and who had not received any excluded concomitant medications through the completion of Part A. Overall number analyzed is the number of participants available for analyses.
Measure: Median (Full Range); unit: hours (h)
Groups:
- Part B: Control Arm: Pevonedistat 10 mg/m^2 + Azacitidine 75 mg/m^2: Participants with normal renal and hepatic function with hematologic malignancies (MDS and AML) who completed Part A and a 4 to 7 days of washout period received pevonedistat 10 mg/m^2, infusion, IV, once, on Days 1, 3, and 5 in each 28-day treatment cycle in combination with azacitidine 75 mg/m^2, injection, SC in Cycle 1 or SC or IV in Cycle 2 and subsequent cycles, once on Day 1 through Day 7 or Day 1 through Day 5, and on Days 8 and 9 until symptomatic deterioration or PD, discontinuation for any reason, study stopped by the sponsor, or up to 12 cycles.
- Part B: Renal Arm: Pevonedistat 10 mg/m^2 + Azacitidine 75 mg/m^2: Participants with severe renal impairment with hematologic malignancies (MDS and AML) who completed Part A and a 4 to 7 days of washout period received pevonedistat 10 mg/m^2, infusion, IV, once, on Days 1, 3, and 5 in each 28-day treatment cycle in combination with azacitidine 75 mg/m^2, injection, SC in Cycle 1 or SC or IV in Cycle 2 and subsequent cycles, once on Day 1 through Day 7 or Day 1 through Day 5, and on Days 8-9 until symptomatic deterioration or PD, discontinuation for any reason, study stopped by the sponsor, or up to 12 cycles.
- Part B: Mild Hepatic Arm: Pevonedistat 10 mg/m^2 + Azacitidine 75 mg/m^2: Participants with mild hepatic impairment with hematologic malignancies (MDS and AML) who completed Part A and a 4 to 7 days of washout period received pevonedistat 10 mg/m^2, infusion, IV, once, on Days 1, 3, and 5 in each 28-day treatment cycle in combination with azacitidine 75 mg/m^2, injection, SC in Cycle 1 or SC or IV in Cycle 2 and subsequent cycles, once on Day 1 through Day 7 or Day 1 through Day 5, and on Days 8-9 until symptomatic deterioration or PD, discontinuation for any reason, study stopped by the sponsor, or up to 12 cycles.
- Part B: Control Arm: Pevonedistat 15 mg/m^2 + Azacitidine 75 mg/m^2: Participants with normal renal and hepatic function with hematologic malignancies (MDS and AML) who completed Part A and a 4 to 7 days of washout period received pevonedistat 15 mg/m^2, infusion, IV, once, on Days 1, 3, and 5 in each 28-day treatment cycle in combination with azacitidine 75 mg/m^2, injection, SC in Cycle 1 or SC or IV in Cycle 2 and subsequent cycles, once on Day 1 through Day 7 or Day 1 through Day 5, and on Days 8 and 9 until symptomatic deterioration or PD, discontinuation for any reason, study stopped by the sponsor, or up to 12 cycles.
- Part B: Renal Arm: Pevonedistat 15 mg/m^2 + Azacitidine 75 mg/m^2: Participants with severe renal impairment with hematologic malignancies (MDS and AML) who completed Part A and a 4 to 7 days of washout period received pevonedistat 15 mg/m^2, infusion, IV, once, on Days 1, 3, and 5 in each 28-day treatment cycle in combination with azacitidine 75 mg/m^2, injection, SC in Cycle 1 or SC or IV in Cycle 2 and subsequent cycles, once on Day 1 through Day 7 or Day 1 through Day 5, and on Days 8-9 until symptomatic deterioration or PD, discontinuation for any reason, study stopped by the sponsor, or up to 12 cycles.
- Part B: Mild Hepatic Arm: Pevonedistat 15 mg/m^2 + Azacitidine 75 mg/m^2: Participants with mild hepatic impairment with hematologic malignancies (MDS and AML) who completed Part A and a 4 to 7 days of washout period received pevonedistat 15 mg/m^2, infusion, IV, once, on Days 1, 3, and 5 in each 28-day treatment cycle in combination with azacitidine 75 mg/m^2, injection, SC in Cycle 1 or SC or IV in Cycle 2 and subsequent cycles, once on Day 1 through Day 7 or Day 1 through Day 5, and on Days 8-9 until symptomatic deterioration or PD, discontinuation for any reason, study stopped by the sponsor, or up to 12 cycles.
- Part B: Control Arm: Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2: Participants with normal renal and hepatic function with hematologic malignancies (MDS and AML) who completed Part A and a 4 to 7 days of washout period received pevonedistat 20 mg/m^2, infusion, IV, once, on Days 1, 3, and 5 in each 28-day treatment cycle in combination with azacitidine 75 mg/m^2, injection, SC in Cycle 1 or SC or IV in Cycle 2 and subsequent cycles, once on Day 1 through Day 7 or Day 1 through Day 5, and on Days 8 and 9 until symptomatic deterioration or PD, discontinuation for any reason, study stopped by the sponsor, or up to 12 cycles.
- Part B: Renal Arm: Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2: Participants with severe renal impairment with hematologic malignancies (MDS and AML) who completed Part A and a 4 to 7 days of washout period received pevonedistat 20 mg/m^2, infusion, IV, once, on Days 1, 3, and 5 in each 28-day treatment cycle in combination with azacitidine 75 mg/m^2, injection, SC in Cycle 1 or SC or IV in Cycle 2 and subsequent cycles, once on Day 1 through Day 7 or Day 1 through Day 5, and on Days 8-9 until symptomatic deterioration or PD, discontinuation for any reason, study stopped by the sponsor, or up to 12 cycles.
- Part B: Mild Hepatic Arm: Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2: Participants with mild hepatic impairment with hematologic malignancies (MDS and AML) who completed Part A and a 4 to 7 days of washout period received pevonedistat 20 mg/m^2, infusion, IV, once, on Days 1, 3, and 5 in each 28-day treatment cycle in combination with azacitidine 75 mg/m^2, injection, SC in Cycle 1 or SC or IV in Cycle 2 and subsequent cycles, once on Day 1 through Day 7 or Day 1 through Day 5, and on Days 8-9 until symptomatic deterioration or PD, discontinuation for any reason, study stopped by the sponsor, or up to 12 cycles.
Arm/Group | Part A: Control Arm: Pevonedistat 20 mg/m^2 | Part A: Renal Arm: Pevonedistat 20 mg/m^2 | Part A: Mild Hepatic Arm: Pevonedistat 20 mg/m^2 | Part B: Control Arm: Pevonedistat 10 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Renal Arm: Pevonedistat 10 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Mild Hepatic Arm: Pevonedistat 10 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Control Arm: Pevonedistat 15 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Renal Arm: Pevonedistat 15 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Mild Hepatic Arm: Pevonedistat 15 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Control Arm: Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Renal Arm: Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Mild Hepatic Arm: Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 10 | 4 | 3 | 0 | 3 | 2 | 0 | 1 | 0 | 10 | 0 | 1
hours (h) | 6.957 [4.25 to 13.88] | 8.493 [7.31 to 10.29] | 9.612 [7.49 to 11.03] |  | 8.795 [7.03 to 9.22] | 10.248 [9.78 to 10.72] |  | 8.98 [8.98 to 8.98] |  | 6.477 [3.93 to 13.37] |  | 6.79 [6.79 to 6.79]

5. Secondary Outcome: Part B: Cmax: Maximum Observed Plasma Concentration for Pevonedistat Following Multiple Dose
Time Frame: Cycle 1 Day 3 pre-dose and at multiple time points (up to 48 hours) post-dose (Cycle length= 28 days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part B: Control Arm: Pevonedistat 10 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Renal Arm: Pevonedistat 10 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Mild Hepatic Arm: Pevonedistat 10 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Control Arm: Pevonedistat 15 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Renal Arm: Pevonedistat 15 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Mild Hepatic Arm: Pevonedistat 15 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Control Arm: Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Renal Arm: Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Mild Hepatic Arm: Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 0 | 3 | 2 | 0 | 1 | 0 | 10 | 0 | 1
ng/mL |  | 74.73 (14.941) | 44.74 (24.579) |  | 128.00 (NA) — Geometric coefficient of variation was not estimable for 1 participant as the values were below the lower limit of quantitation (LLOQ) of the bioanalytical assay. |  | 141.55 (37.468) |  | 75.80 (NA) — Geometric coefficient of variation was not estimable for 1 participant as the values were below the LLOQ of the bioanalytical assay.

6. Secondary Outcome: Parts A, fu: Fraction of Unbound Drug in Plasma for Pevonedistat
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of plasma fraction unbound
Arm/Group | Part A: Control Arm: Pevonedistat 20 mg/m^2 | Part A: Renal Arm: Pevonedistat 20 mg/m^2 | Part A: Mild Hepatic Arm: Pevonedistat 20 mg/m^2
Number analyzed (Participants) | 10 | 4 | 2
percentage of plasma fraction unbound | 5.800 (18.2880) | 7.073 (12.2269) | 5.529 (2.0462)

7. Secondary Outcome: Part B, Cmax: Maximum Observed Plasma Concentration for Azacitidine Following Multiple Dose
Time Frame: Cycle 1 Day 3 pre-dose and at multiple time points (up to 7 hours) post-dose (Cycle length= 28 days)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part B: Control Arm: Pevonedistat 20 milligram per square meter (mg/m^2), infusion, intravenously (IV), once, on Day 1 of Part A in participants with hematologic malignancies, followed by a washout period of approximately 4 to 7 days. Following Part A participants received azacitidine 75 mg/m^2, injection, subcutaneously (SC) in Cycle 1 or SC or IV in Cycle 2 and subsequent cycles, once on Day 1 through Day 7 or Day 1 through Day 5, and on Days 8 and 9 in combination with pevonedistat 20 mg/m^2, infusion, IV, once, on Days 1, 3, and 5 in each 28-day treatment cycle in participants with hematologic malignancies in Part B until symptomatic deterioration or PD, discontinuation for any reason, study stopped by the sponsor, or up to 12 cycles.
- Part B: Renal Arm: Pevonedistat 20 mg/m^2, infusion, intravenously, once, on Day 1 of Part A in participants with hematologic malignancies, followed by a washout period of approximately 4 to 7 days. Following Part A participants received azacitidine 75 mg/m^2, injection, subcutaneously in Cycle 1 or subcutaneously or intravenously in Cycle 2 and subsequent cycles, once on Day 1 through Day 7 or Day 1 through Day 5, and on Days 8-9 in combination with a starting dose of pevonedistat 10 mg/m^2 to a maximum dose of pevonedistat 15 mg/m^2, infusion, intravenously, once, on Days 1, 3, and 5 in each 28-day treatment cycle in participants with hematologic malignancies in Part B until symptomatic deterioration or PD, discontinuation for any reason, study stopped by the sponsor, or up to 12 cycles.
- Part B: Mild Hepatic Arm: Pevonedistat 20 mg/m^2, infusion, intravenously, once, on Day 1 of Part A in participants with hematologic malignancies, followed by a washout period of approximately 4 to 7 days. Following Part A participants received azacitidine 75 mg/m^2, injection, subcutaneously in Cycle 1 or subcutaneously or intravenously in Cycle 2 and subsequent cycles, once on Day 1 through Day 7 or Day 1 through Day 5, and on Days 8 and 9 in combination with a starting dose of pevonedistat 10 mg/m^2 to a maximum dose of pevonedistat 20 mg/m^2, infusion, intravenously, once, on Days 1, 3, and 5 in each 28-day treatment cycle in participants with hematologic malignancies until symptomatic deterioration or PD, discontinuation for any reason, study stopped by the sponsor, or up to 12 cycles.
Arm/Group | Part B: Control Arm | Part B: Renal Arm | Part B: Mild Hepatic Arm
Number analyzed (Participants) | 10 | 4 | 3
ng/mL | 645.4 (34.40) | 918.6 (98.14) | 834.8 (38.23)

8. Secondary Outcome: Part B, Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Azacitidine Following Multiple Dose
Time Frame: Cycle 1 Day 3 pre-dose and at multiple time points (up to 7 hours) post-dose (Cycle length= 28 days)
Population: as for outcome 2
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Part B: Control Arm | Part B: Renal Arm | Part B: Mild Hepatic Arm
Number analyzed (Participants) | 10 | 4 | 3
hours (h) | 0.325 [0.08 to 0.75] | 0.500 [0.32 to 0.53] | 0.250 [0.12 to 0.75]

9. Secondary Outcome: Part B, t1/2z: Terminal Disposition Phase Half-life for Azacitidine Following Multiple-dose
Time Frame: Cycle 1 Day 3 pre-dose and at multiple time points (up to 7 hours) post-dose (Cycle length= 28 days)
Population: as for outcome 2
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Part B: Control Arm | Part B: Renal Arm | Part B: Mild Hepatic Arm
Number analyzed (Participants) | 10 | 4 | 3
hours (h) | 0.706 [0.57 to 1.47] | 1.020 [0.79 to 1.76] | 0.694 [0.67 to 1.13]

10. Secondary Outcome: Part B, AUCτ: Area Under the Concentration-time Curve From Time Zero to the End of the Dosing Interval for Pevonedistat Following Multiple Dose
Time Frame: Cycle 1 Day 3 pre-dose and at multiple time points (up to 48 hours) post-dose (Cycle length= 28 days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part B: Control Arm: Pevonedistat 10 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Renal Arm: Pevonedistat 10 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Mild Hepatic Arm: Pevonedistat 10 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Control Arm: Pevonedistat 15 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Renal Arm: Pevonedistat 15 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Mild Hepatic Arm: Pevonedistat 15 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Control Arm: Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Renal Arm: Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Mild Hepatic Arm: Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 0 | 3 | 2 | 0 | 1 | 0 | 10 | 0 | 1
h*ng/mL |  | 574.168 (19.6797) | 396.240 (14.4663) |  | 884.974 (NA) — Geometric coefficient of variation was not estimable for 1 participant as the values were below the LLOQ of the bioanalytical assay. |  | 848.866 (25.6831) |  | 431.699 (NA) — Geometric coefficient of variation was not estimable for 1 participant as the values were below the LLOQ of the bioanalytical assay.

11. Secondary Outcome: Part B, AUCτ: Area Under the Concentration-time Curve From Time Zero to the End of the Dosing Interval for Azacitidine Following Multiple Dose
Time Frame: Cycle 1 Day 3 pre-dose and at multiple time points (up to 7 hours) post-dose (Cycle length= 28 days)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Part B: Control Arm: Pevonedistat 20 mg/m^2, infusion, IV, once, on Day 1 of Part A in participants with hematologic malignancies, followed by a washout period of approximately 4 to 7 days. Following Part A participants received azacitidine 75 mg/m^2, injection, subcutaneously (SC) in Cycle 1 or SC or IV in Cycle 2 and subsequent cycles, once on Day 1 through Day 7 or Day 1 through Day 5, and on Days 8 and 9 in combination with pevonedistat 20 mg/m^2, infusion, IV, once, on Days 1, 3, and 5 in each 28-day treatment cycle in participants with hematologic malignancies in Part B until symptomatic deterioration or PD, discontinuation for any reason, study stopped by the sponsor, or up to 12 cycles.
Arm/Group | Part B: Control Arm | Part B: Renal Arm | Part B: Mild Hepatic Arm
Number analyzed (Participants) | 10 | 4 | 3
h*ng/mL | 822.457 (31.1338) | 1331.654 (63.1278) | 751.448 (35.3760)

12. Secondary Outcome: Parts A and B, CL: Total Clearance for Pevonedistat
Time Frame: Part A: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose; Part B: Cycle 1 Day 3 pre-dose and at multiple time points (up to 48 hours) post-dose (Cycle length is 28 Days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour (L/h)
Arm/Group | Part A: Control Arm: Pevonedistat 20 mg/m^2 | Part A: Renal Arm: Pevonedistat 20 mg/m^2 | Part A: Mild Hepatic Arm: Pevonedistat 20 mg/m^2 | Part B: Control Arm: Pevonedistat 10 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Renal Arm: Pevonedistat 10 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Mild Hepatic Arm: Pevonedistat 10 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Control Arm: Pevonedistat 15 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Renal Arm: Pevonedistat 15 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Mild Hepatic Arm: Pevonedistat 15 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Control Arm: Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Renal Arm: Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Mild Hepatic Arm: Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 10 | 4 | 3 | 0 | 3 | 2 | 0 | 1 | 0 | 10 | 0 | 1
liters per hour (L/h) | 32.149 (64.5489) | 29.167 (31.5125) | 34.476 (56.9322) |  | 32.721 (36.0104) | 51.628 (9.1794) |  | 32.361 (NA) — Geometric coefficient of variation was not estimable for 1 participant as the values were below the LLOQ of the bioanalytical assay. |  | 44.259 (24.9426) |  | 65.746 (NA) — Geometric coefficient of variation was not estimable for 1 participant as the values were below the LLOQ of the bioanalytical assay.

13. Secondary Outcome: Part B, CL/F: Apparent Clearance for Azacitidine
Time Frame: Cycle 1 Day 3 pre-dose and at multiple time points (up to 8 hours) post-dose (Cycle length= 28 days)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Part B: Control Arm | Part B: Renal Arm | Part B: Mild Hepatic Arm
Number analyzed (Participants) | 10 | 4 | 3
L/h | 171.301 (34.6321) | 106.238 (74.8634) | 180.744 (21.1071)

14. Secondary Outcome: Part B, CLR: Renal Clearance for Pevonedistat
Time Frame: Cycle 1 Day 3 pre-dose and at multiple time points (up to 8 hours) post-dose (Cycle length= 28 days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Part B: Control Arm: Pevonedistat 10 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Renal Arm: Pevonedistat 10 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Mild Hepatic Arm: Pevonedistat 10 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Control Arm: Pevonedistat 15 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Renal Arm: Pevonedistat 15 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Mild Hepatic Arm: Pevonedistat 15 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Control Arm: Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Renal Arm: Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Mild Hepatic Arm: Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 0 | 2 | 2 | 0 | 1 | 0 | 10 | 0 | 1
L/h |  | 0.298 (51.0558) | 0.492 (36.0553) |  | 0.069 (NA) — Geometric coefficient of variation was not estimable for 1 participant as the values were below the LLOQ of the bioanalytical assay. |  | 0.516 (147.7469) |  | 0.062 (NA) — Geometric coefficient of variation was not estimable for 1 participant as the values were below the LLOQ of the bioanalytical assay.

15. Secondary Outcome: Part B, CLR: Renal Clearance for Azacitidine
Time Frame: Cycle 1 Day 3 pre-dose and at multiple time points (up to 8 hours) post-dose (Cycle length= 28 days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Part B: Control Arm | Part B: Renal Arm | Part B: Mild Hepatic Arm
Number analyzed (Participants) | 10 | 3 | 3
L/h | 0.909 (134.3959) | 0.161 (207.8515) | 0.445 (167.4353)

16. Secondary Outcome: Parts A and B, Vss: Volume of Distribution at Steady-state of Pevonedistat
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)
Arm/Group | Part A: Control Arm: Pevonedistat 20 mg/m^2 | Part A: Renal Arm: Pevonedistat 20 mg/m^2 | Part A: Mild Hepatic Arm: Pevonedistat 20 mg/m^2 | Part B: Control Arm: Pevonedistat 10 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Renal Arm: Pevonedistat 10 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Mild Hepatic Arm: Pevonedistat 10 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Control Arm: Pevonedistat 15 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Renal Arm: Pevonedistat 15 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Mild Hepatic Arm: Pevonedistat 15 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Control Arm: Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Renal Arm: Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2 | Part B: Mild Hepatic Arm: Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 10 | 4 | 3 | 0 | 3 | 2 | 0 | 1 | 0 | 10 | 0 | 1
Liters (L) | 219.288 (124.3584) | 293.614 (36.3707) | 353.570 (55.0197) |  | 351.749 (23.5066) | 729.013 (3.2642) |  | 336.922 (NA) — Geometric coefficient of variation was not estimable for 1 participant as the values were below the LLOQ of the bioanalytical assay. |  | 370.563 (44.2326) |  | 573.044 (NA) — Geometric coefficient of variation was not estimable for 1 participant as the values were below the LLOQ of the bioanalytical assay.

17. Secondary Outcome: Part B, Vz/F: Apparent Volume of Distribution of Azacitidine
Time Frame: Cycle 1 Day 3 pre-dose and at multiple time points (up to 8 hours) post-dose (Cycle length= 28 days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Part B: Control Arm | Part B: Renal Arm | Part B: Mild Hepatic Arm
Number analyzed (Participants) | 10 | 4 | 3
L | 190.871 (60.0093) | 167.610 (92.9284) | 211.139 (8.4099)

18. Secondary Outcome: Part B: Percentage of AML Participants With Complete Response/ Remission (CR) or CR With Incomplete Blood Count Recovery (CRi) or Partial Response (PR)
Description: Disease response in AML are based on international working group (IWG) for diagnosis, standardization of response criteria, treatment outcomes, and reporting standards for therapeutic trials in AML. For AML participants, all CR includes both CR and CRi. CR: morphologic leukemia-free state with absolute neutrophil count (ANC) of greater than (>) 1000 per microliter (/mcL) and platelets of greater than or equal to (>=) 100,000/mcL, and no residual evidence of extramedullary leukemia. CRi: After chemotherapy, some participants fulfill all criteria for CR except for residual neutropenia (less than [<] 1000/mcL) or thrombocytopenia (<100,000/mcL). PR: requires all hematologic values for a CR but with a decrease of at least 50 percent (%) in the percentage of blasts to 5% to 25% in the bone marrow aspirate. A value of less than or equal to (<=) 5% blasts may also be considered a PR if Auer rods are present.
Time Frame: Cycle 2 Day 22, Cycles 5, 8, and 11 (between Days 15 and 28), and every 6 cycles (up to 2 years 9 months) (Cycle length= 28 days)
Population: Response-evaluable population included participants who received at least 1 dose of study drug, had a baseline disease assessment, and had at least 1 postbaseline disease assessment to analyze response. Percentages are rounded off to whole number at the nearest decimal.
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Control Arm | Part B: Renal Arm | Part B: Mild Hepatic Arm
Number analyzed (Participants) | 8 | 1 | 2
percentage of participants
  CR or CRi | 13 | 0 | 0
  PR | 0 | 0 | 0

19. Secondary Outcome: Part B: Percentage of MDS and CMML Participants With CR, PR or Hematologic Improvement (HI)
Description: Disease response in MDS and CMML was based on best overall response (CR+PR+HI) as determined by investigator using revised IWG response criteria for MDS and CMML. CR: morphologic leukemia-free state with absolute neutrophil count (ANC) of greater than (>) 1000 per microliter (/mcL) and platelets of greater than or equal to (>=) 100,000/mcL, and no residual evidence of extramedullary leukemia. PR: requires all hematologic values for a CR but with a decrease of at least 50 percent (%) in the percentage of blasts to 5% to 25% in the bone marrow aspirate. A value of less than or equal to (<=) 5% blasts may also be considered a PR if Auer rods are present. HI: erythropoietic (HI-E): Hemoglobin increase of ≥ 1.5 g/dL untransfused, for red blood cells (RBC) transfusions performed for hemoglobin ≤ 9.0: reduction in RBC units transfused in 8 weeks by ≥ 4 units compared to the number of units transfused in the 8 weeks prior to treatment. No participants with CMML were enrolled in this study.
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Control Arm | Part B: Renal Arm | Part B: Mild Hepatic Arm
Number analyzed (Participants) | 8 | 1 | 2
percentage of participants
  MDS CR | 38 | 0 | 0
  MDS PR | 0 | 0 | 0
  MDS HI | 0 | 0 | 0

20. Secondary Outcome: Part B: Percentage of HR MDS and AML Participants With Overall Response
Description: Overall Response Rate is defined as CR+CRi+PR+HI. CR:≤5% myeloblasts with normal maturation of all bone marrow(BM)cell lines,≥11g/dL Hgb,≥100*10^9/L pl,≥1.0*10^9/L neutrophils,0% blasts in peripheral blood;PR:all CR criteria met except BM blasts ≥50% decrease over pretreatment but still >5%;HI:Hgb increase(inc) ≥1.5g/dL if baseline(BL)<11 g/dL;pl inc≥30*10^9/L if BL>20*10^9/L or inc from <20*10^9/L to >20*10^9/L and by 100%;neutrophil inc by 100%;absolute inc of >0.5*10^9/L if BL<100*10^9/L.For AML-CR:morphologic leukemia-free state >1.0*10^9 neutrophils,≥100*10^9/L pl,transfusion independence,no residual evidence of extramedullary leukemia;CR with incomplete blood count recovery:fulfill CR criteria except residual neutropenia (<1000/μL) or thrombocytopenia (<100,000/μL);PR:all CR hematological values but ≥50% decrease in BM aspirate.
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Control Arm | Part B: Renal Arm | Part B: Mild Hepatic Arm
Number analyzed (Participants) | 8 | 1 | 2
percentage of participants | 50 | 0 | 0

21. Secondary Outcome: Part B: Duration of CR, PR and HI
Description: Duration of response in participants with disease response (CR+PR+HI) for hematologic malignancies is time between first documentation of response and disease progression. Duration of response will be determined by the investigator using the revised IWG response criteria.
Time Frame: From first documentation of response up to disease progression (up to 2 years 9 months)
Population: Response-evaluable population included participants who received at least 1 dose of study drug, had a baseline disease assessment, and had at least 1 postbaseline disease assessment to analyze response. Overall number of participants analyzed is the number of participants with disease response (CR+PR+HI) for hematologic malignancies.
Measure: Median (Full Range); unit: days
Arm/Group | Part B: Control Arm | Part B: Renal Arm | Part B: Mild Hepatic Arm
Number analyzed (Participants) | 4 | 0 | 0
days | NA [NA to NA] — Data for median and full range was not estimable due to insufficient number of participants with events (i.e., disease progression). |  |

22. Secondary Outcome: Part B: Percentage of Solid Tumors Participants With CR or PR
Description: Disease response in solid tumors was based on best overall response (CR+PR) as determined by investigator using the RECIST version 1.1 criteria. CR: disappearance of all target lesions with any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to <10 millimeter (mm) and disappearance of all nontarget lesions and normalization of tumor marker level with all lymph nodes must be nonpathological in size (<10 mm short axis); PR: At least a 30% decrease from baseline in the sum of diameters of target lesions, taking as reference the baseline sum of diameters and Persistence of one or more nontarget lesion(s) or/and maintenance of tumor marker level above the normal limits. No participants with solid tumors were enrolled in this study.
Time Frame: as for outcome 18
Population: No participants with solid tumors were enrolled in this study.
Arm/Group | Part B: Control Arm | Part B: Renal Arm | Part B: Mild Hepatic Arm
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the study start up to end of study (up to approximately 2 years 9 months)
Description: At each visit investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by participant or observed by investigator was recorded, irrespective of relation to study treatment. Safety population included all participants who received at least 1 dose of study drug. As pre-specified in protocol and SAP, data for adverse events are reported separately for Part A and Part B based on their renal and/or hepatic function.
Groups:
- Part A: Control Arm: Pevonedistat 20 milligram per square meter (mg/m^2), infusion, intravenously (IV), once, on Day 1 of Part A in participants with hematologic malignancies, followed by a washout period of approximately 4 to 7 days.
- Part A: Renal Arm: Pevonedistat 20 mg/m^2, infusion, intravenously, once, on Day 1 of Part A in participants with renal hematologic malignancies, followed by a washout period of approximately 4 to 7 days.
- Part A: Mild Hepatic Arm: Pevonedistat 20 mg/m^2, infusion, intravenously, once, on Day 1 of Part A in participants with mild hematologic malignancies, followed by a washout period of approximately 4 to 7 days.
- Part B: Control Arm: Following Part A participants received azacitidine 75 mg/m^2, injection, subcutaneously (SC) in Cycle 1 or SC or IV in Cycle 2 and subsequent cycles, once on Day 1 through Day 7 or Day 1 through Day 5, and on Days 8 and 9 in combination with pevonedistat 20 mg/m^2, infusion, IV, once, on Days 1, 3, and 5 in each 28-day treatment cycle in participants with hematologic malignancies in Part B until symptomatic deterioration or PD, discontinuation for any reason, study stopped by the sponsor, or up to 12 cycles.
- Part B: Renal Arm: Following Part A participants received azacitidine 75 mg/m^2, injection, subcutaneously in Cycle 1 or subcutaneously or intravenously in Cycle 2 and subsequent cycles, once on Day 1 through Day 7 or Day 1 through Day 5, and on Days 8-9 in combination with a starting dose of pevonedistat 10 mg/m^2 to a maximum dose of pevonedistat 15 mg/m^2, infusion, intravenously, once, on Days 1, 3, and 5 in each 28-day treatment cycle in participants with renal hematologic malignancies in Part B until symptomatic deterioration or PD, discontinuation for any reason, study stopped by the sponsor, or up to 12 cycles.
- Part B: Mild Hepatic Arm: Following Part A participants received azacitidine 75 mg/m^2, injection, subcutaneously in Cycle 1 or subcutaneously or intravenously in Cycle 2 and subsequent cycles, once on Day 1 through Day 7 or Day 1 through Day 5, and on Days 8 and 9 in combination with a starting dose of pevonedistat 10 mg/m^2 to a maximum dose of pevonedistat 20 mg/m^2, infusion, intravenously, once, on Days 1, 3, and 5 in each 28-day treatment cycle in participants with mild hematologic malignancies in Part B until symptomatic deterioration or PD, discontinuation for any reason, study stopped by the sponsor, or up to 12 cycles.
Arm/Group | Part A: Control Arm | Part A: Renal Arm | Part A: Mild Hepatic Arm | Part B: Control Arm | Part B: Renal Arm | Part B: Mild Hepatic Arm
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/4 | 0/3 | 2/10 | 2/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/4 | 0/3 | 7/10 | 3/4 | 2/3
Other Adverse Events (participants affected / at risk) | 2/10 | 1/4 | 1/3 | 10/10 | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Control Arm (N=10) | Part A: Renal Arm (N=4) | Part A: Mild Hepatic Arm (N=3) | Part B: Control Arm (N=10) | Part B: Renal Arm (N=4) | Part B: Mild Hepatic Arm (N=3)
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia pseudomonal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Thyroid gland abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Control Arm (N=10) | Part A: Renal Arm (N=4) | Part A: Mild Hepatic Arm (N=3) | Part B: Control Arm (N=10) | Part B: Renal Arm (N=4) | Part B: Mild Hepatic Arm (N=3)
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 2 | 0
Anal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 3 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Blast cell count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 2
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 3 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Bullous haemorrhagic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Catheter site haematoma (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 2 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 4 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 4 | 2 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 2 | 0 | 0
Injection site nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Injection site pain (General disorders) | 0 | 0 | 0 | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Leukostasis syndrome (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lip blister (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lip ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 2 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1 | 1 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oral purpura (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 0
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 6 | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Urethral haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0 | 4 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT03814005/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-23): https://cdn.clinicaltrials.gov/large-docs/05/NCT03814005/SAP_001.pdf